CLINICAL TRIAL: NCT02417909
Title: Quality of Life and Psychological Difficulties in Relation With the Weight of Teenagers
Brief Title: Overweight, Quality of Life and Psychological Difficulties in Teenagers
Acronym: QOL-ADOB
Status: Completed | Type: Observational
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Other Study IDs: RC-P0011
Record Dates: First submitted 2015-04-13; First posted 2015-04-16 (Estimated); Last update posted 2015-08-05 (Estimated); Status verified 2015-05

CONDITIONS: Obesity
Keywords: Obesity; quality of life; teenagers; psychological impact
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy volunteers: This group is composed of healthy teenagers that volunteered to participate in the trial and that will answer questionnaires about quality of life. Parents will anwser questionnaires too.
  Interventions: Other: questionnaires about quality of life
- Obese teenagers: This group is composed of obese teenagers that have been recruited to participate in the trial and that will answer different questionnaires quality of life. Parents will anwser questionnaires too.
  Interventions: Other: questionnaires about quality of life

INTERVENTIONS:
Other: questionnaires about quality of life — all teenagers included in the trial and their parents must complete the questionnaires given of them the day of enrollment.

SUMMARY:
Obesity is a major public heath issue. It may have various impacts on a patient's life by causing psychological problems, altering a patient's quality of life,etc. These led to the investigators' hypothesis which is examining the psychological dimensions of a teenager suffering for obesity.

DETAILED DESCRIPTION:
There are two groups in this study : healthy volunteers and teenagers suffering from obesity.

Patients and healthy volunteers will come to the nutrition clinic center Naturalpha where the patient will complete a questionnaire. The included patients will also complete a questionnaire privately (without the presence of the parents), they will also be weighted and measured.

No further tests or questionnaires will be given after the enrollment day.

ELIGIBILITY:
Inclusion Criteria for obese teenagers :

* Patients aged between 11 and 16 years old at the moment of enrollment.
* Body Mass Index between the 1st and 2nd degree of the obesity zone (over the 97th percentile curve regarding corpulence curves of the Plan National Nutrition Santé (PNNS) based on the gender (boys/girls))
* The teenagers have an appointment in the pediatric unit of the Saint Vincent de Paul Hospital for an examination regarding excess weight

Inclusion Criteria for average weighted teenagers :

* Patients aged between 11 and 16 years old at the moment of enrollment
* Body Mass Index located between the 3rd and the 97th percentile on the corpulence curves of the PNNS
* The teenagers and their parents have replied to and advertisement of the trial

Exclusion Criteria for obese children :

* Body Mass Index over the 97th percentile curve on the corpulence curves of the PNNS
* Handicapped teenagers

Exclusion Criteria for average weighted children :

* Body Mass Index over the 97th percentile curve or under the 3rd percentile curve on the corpulence curves of the PNNS
* Handicapped, asthmatic, obese or diabetic teenagers

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Two categories of teenagers will be included : obese teenagers and average weighted volonteers
Sampling Method: Non-Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2011-07; Primary Completion 2015-01 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Compare the quality of life of obese and average weighted teenagers | day of enrollment
  patients are weighted, measured and are asked to complete quality of life questionnaires. The parents are also asked to complete a questionnaire.
  The questionnaires answered by the teenagers are KIDSCREEN; CES-D; STAI-C; PJNA; EPADV; EPCDV and EQRI, they will be analysed along with the questionnaires completed by the parents, inorder to compare the quality of life of obese and average weighted teenagers.

SECONDARY OUTCOMES:
Compare psychopathologic symptoms (depression, anxiety and social anxiety) in both populations | day of enrollement
  Patients are asked to complete quality of life questionnaires. The parents are also asked to complete a questionnaire.
Compare the satisfaction of the needs described in the theory of auto-determination in both populations | day fo enrollment
  Patients are asked to complete quality of life questionnaires. The parents are also asked to complete a questionnaire.
Explore the link between endured stigmatisation and self esteem for obese teenagers | day of enrollment
  Patients are asked to complete quality of life questionnaires. The parents are also asked to complete a questionnaire.
Explore the effect of the support of the needs described in the auto-determination theory and their link to endured stigmatisation, quality of life and self esteem, for obese teenagers. | day of enrollment
  Patients are asked to complete quality of life questionnaires. The parents are also asked to complete a questionnaire.
Explore the possible links between the measured concepts | day of enrollment
  Patients are asked to complete quality of life questionnaires. The parents are also asked to complete a questionnaire. These questionnaires will then be analysed in order to check for possible links between the secondary outcome measures wirtten above.

CONTACTS AND LOCATIONS:
Overall Officials: Gronnier Pascale, MD, Principal Investigator — Groupment des Hôpitaux de l'Institut Catholique de Lille; Gueorguieva Iva, MD, Principal Investigator — Centre Hospitalier Universitaire de Lille